CLINICAL TRIAL: NCT05489510
Title: Safety and Effectiveness of the PXL-Platinum 330 System for Corneal Collagen Cross-Linking in Eyes With Corneal Thinning Conditions
Brief Title: PXL-Platinum 330 in Eyes With Corneal Thinning Conditions
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Vishal Jhanji (Other)
Responsible Party: Sponsor-Investigator, Vishal Jhanji, Professor of Ophthalmology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY21040139
Record Dates: First submitted 2022-03-10; First posted 2022-08-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Corneal Thinning; Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Heart Rate

STUDY DESIGN:
Intervention Model Description: Prospective, double-arm, randomized single-site study
Who Masked: Investigator
Masking Description: Subjects will be assigned randomly to either pulsed or continuous lighting.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Pulsed lighting (Other)
  Interventions: Combination Product: Pulsed or continuous lighting
- Continuous lighting (Other)
  Interventions: Combination Product: Pulsed or continuous lighting

INTERVENTIONS:
Combination Product: Pulsed or continuous lighting — The cross-linking procedures will be performed on an outpatient basis using the PXL Platinum 330 System (UVA light source and riboflavin solution).

SUMMARY:
This study is being conducted to evaluate the safety and effectiveness of using the PXL Platinum 330 system for performing corneal collagen cross-linking (CXL) for the treatment of corneal thinning disorders. The PXL Platinum 330 system is a combination product consisting of a UVA 365 nm wavelength light source (PXL Platinum 330 Illumination System) and riboflavin (Peschke-TE 0.25% ophthalmic solution or Peschke-L 0.23% ophthalmic solution) administered in conjunction with the UVA light as a photosensitizer.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and effectiveness of corneal collagen cross-linking (performed using the PXL-Platinum 330 system) for treating corneal curvature and biomechanical anomalies associated with corneal thinning conditions, e.g., progressive or non-progressive keratoconus, pellucid marginal degeneration, and treatment of patients with bacterial or fungal keratitis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Presence of central or inferior steepening.
* Axial topography consistent with keratoconus, post-surgical ectasia, or pellucid marginal degeneration.
* Presence of one or more findings associated with keratoconus or pellucid marginal degeneration, such as: a. Fleischer ring b. Vogt's striae c. Decentered corneal apex d. Munson's sign e. Rizzutti's sign f. Apical Corneal scarring consistent with Bowman's breaks g. Scissoring of the retinoscopic reflex h. Crab-claw appearance on topography
* Steepest keratometry (Kmax) value ≥ 47.20 D.
* I-S keratometry difference > 1.5 D on the Pentacam/Galilei/Orbscan/Cassini map or topography map.
* Posterior corneal elevation >16 microns.
* Thinnest corneal point <485 microns.
* Predicted Post LASIK/PRK stromal ablation depth <350 microns or expected keratometry >47.2 D, or patients undergoing PRK/SMILE in keratoconus suspect eye.s 10. Bacterial or fungal corneal keratitis persistent and not responding despite > 2 weeks of standard antimicrobial therapy or with rapid. progression of corneal thinning, with loss of >25% corneal thickness
* Contact Lens Wearers Only: a. Removal of contact lenses for the required period of time prior to the screening refraction: Contact Lens Type Minimum Discontinuation Time Soft 1 Week Soft Extended Wear 2 Weeks Soft Toric 3 Weeks Rigid gas permeable 2 Weeks per decade of wear
* Signed written informed consent.
* Willingness and ability to comply with schedule for follow-up.

Exclusion Criteria:

* Eyes classified as either normal or atypical normal on the severity grading scheme.
* Corneal pachymetry at the screening exam that is <300 microns at the thinnest point in the eye(s) to be treated.
* Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications, for example:

  1. History of or active corneal disease (e.g., herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, acanthomeoeba, etc.)
  2. Clinically significant corneal scarring in the CXL treatment zone that is not related to keratoconus or, in the investigator's opinion, will interfere with the cross-linking procedure.
* Pregnancy (including plan to become pregnant) or lactation during the course of the study.
* A known sensitivity to study medications.
* Patients with nystagmus or any other condition that would prevent a steady gaze during the CXL treatment or other diagnostic tests.
* Patients with a current condition that, in the physician's opinion, would interfere with or prolong epithelial healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
PXL-Platinum 330 system | 12 months
  Keratometry

OTHER OUTCOMES:
Efficacy measurements by best spectacle-corrected visual acuity | 12 months
  Percentage of eyes that had a BSCVA worse than 20/40

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Jhanji, MD, Principal Investigator — UPMC Eye Center
Locations (1):
- UPMC Eye Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
In addition to UPMC having access to identifiable information, Peschke Meditrade of Switzerland will have access to de-identifiable information.
Supporting Information: SAP
Time Frame: An indefinite period.
Access Criteria: Deidentified individual participant data sets with other researchers outside of your study team.